CLINICAL TRIAL: NCT06926205
Title: CHOP Plus Mosunetuzumab as First Line in Patients With Richter´s Syndrome: a Phase II Study of the Spanish Group of CLL
Acronym: GELLC9RICHTER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GELLC (Grupo Español de Leucemia Linfocítica Crónica) (Other)
Collaborators: Evidenze Health España (CRO) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELLC-9-RICHTER/M043880; 2023-505621-13-00 (EU CTIS Number); NCT06521996 (obsolete NCT alias)
Record Dates: First submitted 2025-03-17; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Richter Syndrome
Keywords: Richter Syndrome

STUDY DESIGN:
Intervention Model Description: 6 cycle of Mosunetuzumab+CHOP and den 11 cycle more of mosunetuzumab on monotherapy to first line of patients with Richter Syndrome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mosunetuzumab (Experimental): 6 cycle of mosunetuzumab+CHOP and then 11 cycles more of Mosunetuzumab on monotherapy.
  Interventions: Drug: Mosunetuzumab (IV)

INTERVENTIONS:
Drug: Mosunetuzumab (IV) — 6 cycle of Mosunetuzumab+CHOP and then 11 cycles more of mosunetuzumab on mnotherapy

SUMMARY:
The goal of this clinical trial is to learn if drug Mosunetuzumab works to treat Richter´syndrome . It will also learn about the safety of drug Mosunetuzumab. The main questions it aims to evaluate the efficacy of mosunetuzumab combined with CHOP (M-CHOP) after the end of induction in patients with Richter´s Syndrome who have never received thearapy

What medical problems do participants have when taking drug Mosunetuzumab? Patients with Richter´s Syndrome

Participants will:

Take drug Mosunetuzumab+CHOP during 6 cycle and they if they are not candidate to Alothasplant continuing 11 cycles more with mosunetuzumab on monoterapy Visit the clinic once every 23weeks for checkups and tests

DETAILED DESCRIPTION:
Patients with Richter´s Syndrome received 6 cycle of Mosunetuzumab+CHOP. At the EoI, in patients achieving stable disease (SD) or in patients with partial response (PR) or complete response (CR) who are not candidates to consolidation with cellular therapy, mosunetuzumab as monotherapy will be administered over eleven 21-day cycles (approximately 10 months) or until disease progression or unacceptable toxicity, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent as described in Section 13.2, which includes compliance with the requirements and restrictions listed in the Informed Consent Form and this protocol.
2. Aged between 18 and 79 years at the time of signing the Informed Consent Form
3. Ability to comply with the study protocol and procedures and required hospitalizations, in the investigator's judgement.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2.
5. Adult patients with previously untreated, histologically proven Richter's syndrome, diffuse large B cell variants, following WHO 2008 criteria (Swerdlow SH, 2008).
6. Screening flow cytometry or immunohistochemistry (IHC) evidence of CD20 positive disease as per central review (dim expression of CD20 is acceptable)
7. Adequate BM function independent of growth factor or transfusion at screening as follows unless cytopenia is clearly due to marrow involvement of CLL:

   1. Platelet count ≥75 x 109/L; in cases of thrombocytopenia clearly due to marrow involvement of CLL (per the discretion of the investigator), platelet count should be ≥ 30 x 109/L.
   2. ANC ≥1 x 109/L unless neutropenia is clearly due to marrow involvement of CLL (per the discretion of the investigator)
   3. Total hemoglobin ≥ 9 g/dL unless anemia is due to marrow involvement of CLL (per the discretion of the investigator)
8. Measured or estimated creatinine clearance ≥ 45 mL/min by institutional standard method.
9. Life expectancy > 3 months
10. For women of childbearing potential (WOCBP): agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year, and agreement to refrain from donating eggs, during the treatment period and for at least 3 months after the last dose of mosunetuzumab and 3 months after the last dose of tocilizumab (if applicable).

    1. It is recommended to remain abstinent or use contraception for 12 months after the final dose of cyclophosphamide, doxorubicin, or vincristine.
    2. A woman is considered to be of childbearing potential (WOCBP) if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
    3. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
    4. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
    5. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the Informed Consent Form.
11. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

    1. With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 60 days after the final dose of tocilizumab (if applicable) and must remain abstinent or use a condom for 12 months after the final dose of cyclophosphamide, doxorubicin, or vincristine to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
    2. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of preventing drug exposure. If required per local guidelines or regulations, information about the reliability of abstinence will be described in the Informed Consent Form.

Exclusion Criteria:

1. Pregnant or breastfeeding or intending to become pregnant during the study or within 3 months after the final dose of mosunetuzumab.

   a) WOCBP must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment. If a serum pregnancy test has not been performed within 14 days prior to receiving first study treatment, a negative urine pregnancy test result (performed within 7 days prior to study treatment) must be available.
2. Participants who have received any of the following treatments prior to study entry:

   a) Treatment with mosunetuzumab or other CD20/CD3-directed bispecific antibodies.
3. Participants who have received any of the following treatments, whether investigational or approved, given to treat RS, within the respective time periods prior to initiation of study treatment:

   1. Autologous SCT within 100 days prior to first mosunetuzumab administration.
   2. Allogeneic stem cell transplant for CLL
   3. CAR T-cell therapy for CLL within 100 days before first study treatment
   4. Systemic corticosteroid treatment ≤ 20 mg/day prednisone or equivalent to control symptoms related to disease progression for a maximum of 5 days before starting C1D1 and inhaled corticosteroids are permitted.
4. Central nervous system (CNS) involvement as documented by spinal fluid cytology or imaging.
5. Transformation of CLL to prolymphocytic leukemia.
6. History of prior malignancy, except for conditions as listed below if patients have recovered from the acute side effects incurred as a result of previous therapy:

   1. Malignancies treated with curative intent and with no known active disease present for ≥ 2 years before enrollment.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated cervical carcinoma in situ without evidence of disease.
   4. Surgically/adequately treated low grade, early stage, localized prostate cancer without evidence of disease.
7. Any of the following laboratory abnormalities:

   1. Calculated creatinine Clearance < 45 mL/min (by institutional standard method.).
   2. Absolute neutrophil count (ANC) < 1.0 x 109/L, unless secondary to bone marrow involvement by CLL.
   3. Platelet count <75 x 109/L except if thrombocytopenia is clearly due to marrow involvement of CLL (per the discretion of the investigator) for which exclusion criteria would be platelet count < 30 x 109/L.
   4. Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetictransaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) >2.5 x upper limit of normal (ULN).
   5. Serum total bilirubin > 1.5 x ULN, except in cases of Gilbert's syndrome.
8. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
9. Contraindication to tocilizumab.
10. Presence of any autoimmune disorder including autoimmune hemolytic anemia or autoimmune thrombocytopenia active at the moment of first dose of therapy.

    a) Participants with a history of disease-related immune thrombocytopenic purpura or autoimmune hemolytic anemia may be eligible.
11. History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Exceptions include the following:

    1. Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
    2. Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    3. Participants with a remote history of, or well-controlled autoimmune disease, with a treatment-free interval from immunosuppressive therapy for 12 months may be eligible after review and discussion with the Coordinators.
12. History of solid organ transplantation
13. Participants with infections requiring IV treatment with antibiotics or hospitalization (Grade 3 or 4) within the last 4 weeks prior to enrollment or known active bacterial, viral (including SARS-CoV-2), fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment.
14. History of confirmed progressive multifocal leukoencephalopathy (PML)
15. Positive serologic HIV test at screening
16. Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology). Participants with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if hepatitis B virus (HBV) DNA is undetectable at the time of screening. These participants must be willing to undergo monthly DNA testing and appropriate prophylactic antiviral therapy as indicated.
17. Acute or chronic hepatitis C virus (HCV) infection. Participants who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation.
18. Known or suspected chronic active Epstein Barr Virus infection (CAEBV).
19. Patients with history of macrophage activation syndrome (MAS)/hemophagocytic lymphohistiocytosis (HLH)
20. Received a live, attenuated vaccine within 4 weeks before first dose of study treatment, or in whom it is anticipated that such a live attenuated vaccine will be required during the study period or within 5 months after the final dose of study treatment.
21. Left ventricular ejection fraction (LVEF) <50% by multiple-gated acquisition (MUGA) scan or echocardiogram.
22. Evidence of any significant, concomitant disease that could affect compliance with the protocol or interpretation of results, including, but not limited to:

    1. significant cardiovascular disease (e.g., New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 3 months, unstable arrhythmia, or unstable angina)
    2. significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
    3. clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis.
    4. current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease.
    5. Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past year and have no residual neurologic deficits as judged by the investigator are allowed.
    6. Participants with a history of epilepsy who have had no seizures in the past 2 years with or without anti-epileptic medications can be eligible.
23. Recent major surgery within 4 weeks prior to first study treatment administration, with the exception of protocol-mandated procedures (e.g., tumor biopsies and bone marrow biopsies)
24. Participants who are in dependence to the Sponsor or an investigator.
25. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes an individual's safe participation in and completion of the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of mosunetuzumab combined with CHOP (M-CHOP) after the end of induction (EoI) in patients with RS who have never received therapy. | During 6 cycles (up to 6 months)
  Primary endpoint will be complete remission (CR) evaluated by an independent review committee according to modified Lugano classification using PET/CT scan (Cheson et al. 2016) after the EoI visit.
  CR is defined as a score of 1, 2 or 3 for lymph nodes and extra-lymphatic sites at PET without new lesions and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. All PET evaluable in patients with at least one dose of mosunetuzumab will be included in the efficacy population.

SECONDARY OUTCOMES:
To evaluate the efficacy of mosunetuzumab combined with CHOP (M-CHOP) after the end of induction (EoI) and maintenance (EoM) in patients with therapy naive RS | During induction ( 6 Cycles- up to 6 months) and manteinace ( 11 cycles more-up to 11 months)
  Evaluated response assesment with CR
To evaluate the efficacy of mosunetuzumab combined with CHOP (M-CHOP) after the end of induction (EoI) and maintenance (EoM) in patients with therapy naive RS | During induction ( 6 Cycles- up to 6 months) and manteinace ( 11 cycles more-up to 11 months)
  Evaluated response assesment with PFS.
To evaluate the efficacy of mosunetuzumab combined with CHOP (M-CHOP) after the end of induction (EoI) and maintenance (EoM) in patients with therapy naive RS | During induction ( 6 Cycles- up to 6 months) and manteinace ( 11 cycles more-up to 11 months)
  Evaluated response assesment with OS
To evaluate the efficacy of mosunetuzumab combined with CHOP (M-CHOP) after the end of induction (EoI) and maintenance (EoM) in patients with therapy naive RS | During induction ( 6 Cycles- up to 6 months) and manteinace ( 11 cycles more-up to 11 months)
  Evaluated response assesment with MRD
To determine the incidence and severity of adverse events. | During induction ( 6 Cycles- up to 6 months) and manteinace ( 11 cycles more-up to11 months)
  Incidence of adverse events (AEs): number and percentage of patients with 1 or more AE.
  Severity of AEs. Treatment duration. Total dose received. Number of cycles and dose modifications. Treatment interruptions and discontinuations
To evaluate the study treatment exposure. | During induction ( 6 Cycles- up to 6 months) and manteinace ( 11 cycles more- up to 11 months)
  Incidence of adverse events (AEs): number and percentage of patients with 1 or more AE.
  Severity of AEs. Treatment duration. Total dose received. Number of cycles and dose modifications. Treatment interruptions and discontinuations

OTHER OUTCOMES:
Biomarkers Objetive: To evaluate the relationship between various screening prognostic markers (clinical and biological) and clinical outcomes | during induction (6 Cycles- up to 6 months) and maintenace ( 11 cycles more- up to 11 months)
  Molecular (IGHV and TP53 status) and genetic prognostic factors (complex karyotype) Clonality MRD response and its relationship with the efficacy outcomes of PFS
Biomarkers Objetive: To evaluate the relationship between various screening prognostic markers (clinical and biological) and clinical outcomes | during induction (6 Cycles- up to 6 months) and maintenace ( 11 cycles more- up to 11 months)
  Molecular (IGHV and TP53 status) and genetic prognostic factors (complex karyotype) Clonality MRD response and its relationship with the efficacy outcomes of OS
Biomarkers Objetives: To assess MRD using several technologies, including ctDNA | During induction ( 6 Cycles- up to 6 months) and manteinace ( 11 cycles more- up to11 months)
  Molecular (IGHV and TP53 status) and genetic prognostic factors (complex karyotype) Clonality MRD response and its relationship with the efficacy outcomes of PFS
Biomarkers Objetives: To assess MRD using several technologies, including ctDNA | During induction ( 6 Cycles- up to 6 months) and manteinace ( 11 cycles more- up to11 months)
  Molecular (IGHV and TP53 status) and genetic prognostic factors (complex karyotype) Clonality MRD response and its relationship with the efficacy outcomes of OS

CONTACTS AND LOCATIONS:
Locations (16):
- Spain (16):
  - Hospital Vall Hebron, Barcelona, Barcelona
  - Hospital Clínic y Porvincial de Barcelona, Barcelona, Barcelona
  - ICO Hospitalet Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - H Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario La Princesa, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Universitario Costa del Sol, Marbella, Málaga
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital de Donostia, Donostia / San Sebastian, San Sebastian
  - Centro Hospitalario Universitario de Santiago, Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario Clínico de Valencia, Valencia, Valencia
  - Hospital Universitario Lozano Blesa, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No
The IPD are property of sponsor of study and not share with any researcher